CLINICAL TRIAL: NCT04026126
Title: Effects of Passive Heat Therapy on Oxygen Consumption and Cardiovascular Fitness in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Paige Geiger, PhD, Professor of Molecular & Integrative Physiology, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00142890; P20GM103418-19 (NIH)
Record Dates: First submitted 2019-06-26; First posted 2019-07-19 (Actual); Results first posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure; Heart Diseases; Cardiovascular Diseases; Endothelial Dysfunction
Keywords: Heat Therapy
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heat Therapy Treatment (Experimental): This study will recruit subjects to participate in heat therapy treatment at the University of Kansas Medical Center (KUMC). After pre-screening, informed consent, and enrollment, all subjects will have baseline hemodynamic assessments as well as VO2max measurements. Subjects will complete 10 heat therapy treatments over the course of 14 days. Hemodynamics will be assessed with the use of the Clearsight© fingertip blood pressure cuff. Within 24-48 hours after the last heat therapy experience, hemodynamic assessments and VO2max will be performed. Blood samples will be collected pre- and post intervention and analyzed for levels of nitric oxide mediators, heat shock protein levels and pro-anti-inflammatory markers.
  Interventions: Behavioral: Heat Therapy Treatment

INTERVENTIONS:
Behavioral: Heat Therapy Treatment — Subjects will undergo 10 hot water immersions of 40.5 degrees Celsius for approximately 45 minutes per session over 14 days. Subjects will be immersed up to the shoulder until rectal temperature reacher 38.5 degrees Celsius (approximately 15-20 minutes). Subjects will then remain in the water bath submerged at waist level to maintain between 38.5 to 39.0 degrees Celsius for another 30 minutes. Following hot water immersion, subjects will be monitored for 10 minutes, or until temperature falls below 38.5 degrees Celsius.

SUMMARY:
The purpose of this study is to determine if enhanced endothelial arterial distensibility observed with heat therapy translates into improved cardiorespiratory fitness. The following aims are proposed: Aim 1: to determine if chronic heat therapy results in improvements in cardiovascular function. Aim 2: To examine potential mechanism(s) of action of heat therapy in cardiovascular function.

DETAILED DESCRIPTION:
The National Institute of Health recognizes heart failure as a major public health problem with a prevalence of over 5.8 million Americans and 23 million people worldwide. Commonly prescribed medications to treat the symptoms associated with this disease are expensive and many are not covered by major health insurance companies. There is a critical need to develop novel treatment and prevention strategies for heart failure. Emerging research highlights the benefits of heat therapy (HT) on metabolic and cardiovascular disease risk. The Geiger laboratory has demonstrated that in obese rats fed a high- fat diet for 12 weeks, weekly HT restored whole body glucose tolerance and skeletal muscle insulin sensitivity. The first comprehensive investigation of long-term HT in young, sedentary humans resulted in improved endothelial function and hemodynamics that were on par with what is typically observed with exercise training in previously sedentary subjects. The purpose of this pilot study is to determine if the enhanced endothelial arterial distensibility observed with HT translates into improved cardiorespiratory fitness. The following aims are proposed:

Aim 1: To determine if chronic HT results in improvements in cardiovascular function. The study team hypothesizes that repeated HT will result in improvement in hemodynamic variables related to arterial distensibility (blood pressure, stroke volume, stroke volume variation, cardiac index and systemic vascular resistance) and that these changes translate to improved cardiovascular function as measured by VO2max.

Aim 2: To examine potential mechanism(s) of action of HT in cardiovascular function. The study team hypothesizes that HT may exerts its beneficial effects via the effect of heat shock proteins (HSPs) on Nitric Oxide (NO) bioavailability. This will be tested by measuring HSPs, NO mediators and inflammatory markers at baseline and post-intervention. There is rapidly growing interest in the use of HT as a global therapeutic approach and alternative or complementary therapy to exercise training for patients with chronic disease. Study findings would be clinically significant as both men and women with higher cardiorespiratory fitness (as indicated by maximal oxygen consumption, VO2max) are at lower risk for cardiovascular disease.

These studies will be the first to examine the ability of chronic heat therapy to increase cardiorespiratory fitness as measured by maximal oxygen consumption, VO2max. These findings could lead to HT as a simple and effective tool for improving cardiovascular health in a variety of populations, particularly those with exercise limitations and comorbid disease states like type 2 diabetes, dementia and cardiovascular disease.

ELIGIBILITY:
Exclusion Criteria:

* Current major cardiovascular disease (i.e.: recent myocardial infarction (heart attack), stroke, angina pectoris, high grade coronary vasculopathy or atherosclerosis, severe valvular disease, cardiac dysrhythmia that requires treatment.
* Current treatment with steroids or immunosuppressive agents
* Cancer
* Serious liver disease
* End-stage renal disease
* Judgement by medical provider that heat therapy poses an undue burden or risk
* Women who are pregnant or plan to become pregnant

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paige C Geiger, Ph.D., Principal Investigator — University of Kansas Medical Center; Brigid Flynn, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited primarily through physician referral; as well as IRB-approved flyers posted at the University of Kansas Medical Center, in the community, and through electronic communications via websites and email. The first participant was enrolled on August 29, 2019 and the last was enrolled on June 24, 2021.
Pre-assignment Details: Of the 15 enrolled participants, all 15 met inclusion criteria and completed treatment.
Groups:
- Heat Therapy Treatment: Participants completed 10 heat therapy treatments (hot water immersions of 40.5 degrees Celsius for approximately 45 minutes per session) over 14 days.
Period: Overall Study
Arm/Group | Heat Therapy Treatment
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 58.6 [50 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15
Weight [Mean (Full Range); unit: kgs] | 80.9 [48 to 120]
Hypertension [Count of Participants; unit: Participants] | 3
Diabetes [Count of Participants; unit: Participants] | 2
Asthma [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Pressure
Description: Systolic and diastolic blood pressure will be monitored using the noninvasive Clearsight (Edward Lifesciences, Irvine, CA) monitor, which incorporates a disposable, single use fingertip cuff.
Time Frame: Blood pressure will be assessed at baseline and 24-48 hours after the last heat therapy session (end of study, ~2.5 weeks after first study visit). As a safety measure only, blood pressure will be monitored during every heat therapy treatment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 15
mmHg
  Systolic Pressure | -2.94 (10.94)
  Diastolic Pressure | 0.85 (4.67)

2. Primary Outcome: Change in Stroke Volume
Description: Stroke volume will be monitored using the noninvasive Clearsight (Edward Lifesciences, Irvine, CA) monitor incorporates a disposable, single use fingertip cuff.
Time Frame: Stroke volume will be assessed at baseline and 24-48 hours after the last heat therapy session (end of study, ~2.5 weeks after first study visit).
Measure: Mean (Standard Deviation); unit: ml/m2
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 15
ml/m2 | 9.02 (268.54)

3. Primary Outcome: Change in Stroke Volume Variation
Description: Stroke volume variation will be monitored using the noninvasive Clearsight (Edward Lifesciences, Irvine, CA) monitor incorporates a disposable, single use fingertip cuff.
Time Frame: Stroke volume variation will be assessed at baseline and 24-48 hours after the last heat therapy session (end of study, ~2.5 weeks after first study visit).
Population: We were unable to collect data on SVV and thus data cannot be reported.
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 0

4. Primary Outcome: Change in Cardiac Index
Description: Cardiac index will be monitored using the noninvasive Clearsight (Edward Lifesciences, Irvine, CA) monitor incorporates a disposable, single use fingertip cuff.
Time Frame: Cardiac index will be assessed at baseline and 24-48 hours after the last heat therapy session (end of study, ~2.5 weeks after first study visit).
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 15
L/min/m^2 | -0.36 (0.51)

5. Primary Outcome: Change in Systemic Vascular Resistance
Description: Systemic vascular resistance will be monitored using the noninvasive Clearsight (Edward Lifesciences, Irvine, CA) monitor incorporates a disposable, single use fingertip cuff.
Time Frame: Systemic vascular resistance will be assessed at baseline and 24-48 hours after the last heat therapy session (end of study, ~2.5 weeks after first study visit).
Measure: Mean (Standard Deviation); unit: dynes/seconds/cm-5
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 15
dynes/seconds/cm-5 | 9.02 (268.54)

6. Primary Outcome: Change in Maximum Oxygen Consumption (VO2max)
Description: Maximum oxygen consumption (VO2max) will be measured using the Bruce Ramp protocol. The Bruce Ramp protocol is a standardized treadmill exercise commonly used in clinical laboratories.
Time Frame: VO2max assessment will be performed at baseline and 24-48 hours after the last heat therapy session (end of study, ~2.5 weeks after first study visit).
Measure: Mean (Standard Deviation); unit: ml/kg/minute
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 15
ml/kg/minute | -0.13 (1.81)

7. Primary Outcome: Change in Concentration of Heat Shock Proteins
Description: Serum levels of heat shock proteins (HSP72, HSP25) and the primary heat shock protein transcription factor (HSF1) will be assessed for change post heat therapy treatment.
Time Frame: Blood analyses will be performed at baseline and 24-48 hours after the last heat therapy session (end of study, ~2.5 weeks after first study visit).
Population: The samples were run for HSP but the data was compromised. The study team were unable to verify study samples and match them to participant IDs. Thus the data was invalid, and there was not enough sample to repeat the analysis.
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 0

8. Primary Outcome: Change in Concentration of Nitric Oxide
Description: Nitric oxide (NO) bioavailability will be assessed for change post heat therapy treatment by measuring nitric oxide and endothelial nitric oxide synthase (eNOS).
Time Frame: as for outcome 7
Population: The samples were run for nitric oxide bioavailability but the data was compromised. The study team were unable to verify study samples and match them to participant IDs. Thus the data was invalid, and there was not enough sample to repeat the analysis.
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 0

9. Primary Outcome: Change in Concentration of Pro/Anti-inflammatory Markers
Description: Pro/anti-inflammatory markers (IL1ra, IL-10, IL-8, IFN, and CRP) will be assessed for change post heat therapy treatment.
Time Frame: as for outcome 7
Population: The samples were run for pro/Anti-inflammatory markers but the data was compromised. The study team were unable to verify study samples and match them to participant IDs. Thus the data was invalid, and there was not enough sample to repeat the analysis.
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data would have been collected between date of enrollment through study completion, approximately 2.5 to 3 weeks.
Arm/Group | Heat Therapy Treatment
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT04026126/Prot_000.pdf